CLINICAL TRIAL: NCT05547334
Title: Effect of Inference Based Approach in Adolescents With OCD
Brief Title: IBA Treatment in Adolescents With OCD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Karakter Kinder- en Jeugdpsychiatrie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 217-22; NL81157.091.22 (Registry Identifier: ToetsingOnline)
Record Dates: First submitted 2022-09-14; First posted 2022-09-21 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Obsessive-Compulsive Disorder in Adolescence

STUDY DESIGN:
Intervention Model Description: A non-concurrent multiple baseline design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A non-concurrent multiple baseline design (Other): A non-concurrent multiple baseline design
  Interventions: Behavioral: Inference Based Approach (IBA)

INTERVENTIONS:
Behavioral: Inference Based Approach (IBA) — The Inference Based Approach (IBA) (as described by Visser et al., 2015 and adapted for use in adolescents by L. Webers)is a focused form of psychotherapy consists of twenty 45-minutes sessions, delivered weekly and carried out as specified in a Dutch session-by-session IBA protocol, containing standardized forms for exercises and homework assignments. Each session has a standard format, starting with agenda setting and evaluating homework assignments, followed by determining and executing a new exercise and determining new homework. The IBA model is based on the assumption that adolescents with OCD and poor inside misjudge the actual state of affairs. It is assumed that certain reasoning processes lead to these erroneous conclusions and distract the childs attention from observable reality.

SUMMARY:
Adolescents with Obsessive-compulsive Disorder (OCD) have obsessions, compulsions or both. OCD is a severe psychiatric disorder, affecting many aspects of the lives of adolescents. The first choice treatment for adolescents with OCD is Cognitive Behavioral Therapy (CBT), consisting of exposure with response prevention (ERP) and cognitive interventions. Considering the substantial group of non-responders to CBT, it is necessary to have more options for effective treatment of OCD. Inference Based Approach (IBA) is already an effective treatment for adults with OCD and is more effective on adults with OCD and poor cognitive insight. It is hypothesized that IBA could be an effective alternative for CBT in treating adolescents with OCD. This study will be a first step in examining the efficacy of IBA as treatment for adolescents with OCD.

The aim of this study is to explore the potential efficacy of IBA as treatment for adolescents with OCD using a non-concurrent multiple baseline design with 8 participants who receive IBA for 20 sessions performed in one psychiatric centre in the Netherlands.

DETAILED DESCRIPTION:
Background of the study:

Adolescents with Obsessive-compulsive Disorder (OCD) have obsessions, compulsions or both (APA, 2014). OCD is a severe psychiatric disorder, affecting many aspects of the lives of adolescents (Weidle et al., 2014; Storch et al., 2018). The first choice treatment for adolescents with OCD is Cognitive Behavioral Therapy (CBT), consisting of exposure with response prevention (ERP) and cognitive interventions (Öst et al., 2016). Treating adolescents with OCD through CBT leads to significant symptom reduction in almost 70% of completed treatments (Öst et al., 2016). However, after completion of treatment, about 50% of adolescents still meet the criteria for OCD (Öst et al., 2016). Adolescents with OCD who do not sufficiently benefit from CBT treatment have severe symptoms, including poor or no insight (Sharma et al., 2021; Nissen & Parner, 2018; Storch et al., 2014). Considering the substantial group of non-responders to CBT, it is necessary to have more options for effective treatment of OCD. Inference Based Approach (IBA) is already an effective treatment for adults with OCD (O'Connor et al., 2005; Visser et al., 2015) and is more effective on adults with OCD and poor cognitive insight (Visser et al., 2015). It is hypothesized that IBA could be an effective alternative for CBT in treating adolescents with OCD. This study will be a first step in examining the efficacy of IBA as treatment for adolescents with OCD.

Objective of the study:

The aim of this study is to explore the potential efficacy of IBA as treatment for adolescents with OCD.

Study design:

A non-concurrent multiple baseline design with 8 participants who receive IBA for 20 sessions perfomed in one psychiatric centre in the Netherlands.

Study population:

8 adolescents from 12 to 17;11 years old with a Diagnostic and Statistical Manual Diploma in Social Medicine (DSM-5) diagnosis of OCD and a total score of 16 or higher on the Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS). All adolescents included in this study completed an evidence-based treatment for OCD prior to participation.

Intervention (if applicable):

20 sessions IBA treatment.

Primary study parameters/outcome of the study:

Severity of OCD, measured with the CY-BOCS;

Secondary study parameters/outcome of the study (if applicable):

OCD symptomatology, measured with three-weekly ratings of the adolescents' obsessions, compulsions and the level of insight.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness (if applicable):

No burden or risks are expected due to specific elements of the IBA intervention used in this study. Contrary to CBT, treatment elements of IBA will not include exposure to feared consequences while trying to not indulge in compulsions. On top of that, obsessions will not be questioned or challenged. These characteristics may help participants stay motivated to complete treatment and experience improvement in OCD-symptoms.

ELIGIBILITY:
In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Primary DSM-5 diagnosis of OCD.
* A total score of 16 or higher on the CY-BOCS.
* Age between 12 and 17;11.
* A completed evidence-based treatment for OCD.
* Medication must be stable for at least one month.

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* No sufficient knowledge of the Dutch language
* Autism spectrum disorder (ASD)**
* Mental retardation (TIQ<80)**
* Acute suicidality (defined as having suicidal thoughts and plans and/or preparations to ending their life)

  * In case of ASD and/or mental retardation, the IBA protocol maybe too challenging. It is expected that the included cognitive elements, specifically when abstract reasoning is asked, will ask too much of these subjects.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in severity of OCD | through study completion, an average of 9 months
  measured with the CY-BOCS at T0 = Study intake (baseline phase);T1 = Start treatment phase; i.e. start IBA treatment; T2 = Post-treatment assessment (after IBA treatment); T3 = Follow-up 3 months post-treatment

SECONDARY OUTCOMES:
Change in OCD symptomatology | three-weekly questions during the intervention
  measured with three-weekly ratings of the adolescents' obsessions, compulsions and the level of insight.
Treatment history (psychotherapy and medication) | T0 = Study intake (baseline phase)
  Treatment history (psychotherapy and medication)
Change in current medication use | through study completion, an average of 9 months
  Current medication use at T0 = Study intake (baseline phase) T1 = Start treatment phase; i.e. start IBA treatment T2 = Post-treatment assessment (after IBA treatment) T3 = Follow-up 3 months post-treatment

IPD SHARING:
Plan to Share IPD: No